CLINICAL TRIAL: NCT05343806
Title: Nifedipine Versus Magnesium Sulfate for Tocolysis in Pregnant Women at 32 - 36 Weeks Gestation With Threatened Preterm Labor
Brief Title: Nifedipine Versus Magnesium Sulfate for Late Preterm Tocolysis
Acronym: ASTOS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Abdallah, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASsiut TOcolytic Study 2
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Threatened Preterm Labor
MeSH Terms: interventions — Nifedipine; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nifedipine (Active Comparator): The initial dose of nifedipine will be 2 × 10 mg nifedipine capsules orally in the first hour, followed by 20 mg slow-release nifedipine every 6 hours for the next 47 hours. In the first hour after starting nifedipine, blood pressure and heart rate will be measured every 15 minutes. If blood pressure remains within the normal limits, treatment will be continued.
  Interventions: Drug: Nifedipine 20 Mg
- Magnesium Sulfate (Active Comparator): Women will receive only MgSo4. A loading dose of MgSo4 will be given immediately after enrollment as 4 gm diluted in 200 mL of saline solution administered intravenous over a period of 20 minutes. Afterwards, the maintenance dose of MgSo4 will be administered intravenous in a dose of 1 gm/hour given as 6 gm diluted in 500 mL saline solution titrated with a rate of 100 mL per hour, then this dose is repeated every 6 hours for 48 hours. Respiratory rate and knee jerk will be assessed hourly for women in the MgSo4 group. Serum magnesium level will be measured if clinically indicated.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Nifedipine 20 Mg — The initial dose of nifedipine will be 2 × 10 mg nifedipine capsules orally in the first hour, followed by 20 mg slow-release nifedipine every 6 hours for the next 47 hours. In the first hour after starting nifedipine, blood pressure and heart rate will be measured every 15 minutes. If blood pressure remains within the normal limits, treatment will be continued.
  Arms: Nifedipine
Drug: Magnesium Sulfate — Women will receive only MgSo4. A loading dose of MgSo4 will be given immediately after enrollment as 4 gm diluted in 200 mL of saline solution administered intravenous over a period of 20 minutes. Afterwards, the maintenance dose of MgSo4 will be administered intravenous in a dose of 1 gm/hour given as 6 gm diluted in 500 mL saline solution titrated with a rate of 100 mL per hour, then this dose is repeated every 6 hours for 48 hours. Respiratory rate and knee jerk will be assessed hourly for women in the MgSo4 group. Serum magnesium level will be measured if clinically indicated.
  Arms: Magnesium Sulfate

SUMMARY:
Objective: This trial is designed to compare between the effectiveness of nifedipine versus magnesium sulfate (MgSO4) for tocolysis in women with threatened preterm labor.

Patient Population: The population will include pregnant women at gestational age between 32 and 36 weeks who are 18 years old or older and have signs of threatened preterm labor.

Study Design: This is a single-center, prospective, randomized controlled clinical trial. A total of 264 women pregnant between 32 and 36 weeks having threatened preterm labor will be enrolled and randomized into two parallel treatment arms. Patients in the group A will receive nifedipine, while patients in group B will MgSO4 only.

Treatment: All patients will be randomized on the day of enrollment. Patients with threatened preterm labor will receive the respective tocolysis in each group. All patients will receive corticosteroids for lung maturity according to the local protocol.

Primary outcome: Number of women not delivered within 48 hours of starting tocolytic therapy.

Secondary outcomes: perinatal mortality, a composite of adverse neonatal outcomes, birth weight, days on ventilation support, length of admission in neonatal intensive care, prolongation of pregnancy more than 7 days, delivery after 37 weeks of gestation, number of days till delivery, maternal mortality, maternal infection, and harm to mother from intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with threatened preterm labor defined as 3 or more uterine contractions in 30 minutes confirmed by cardiotocography.
2. Gestational age from 32 week + 0 days to (inclusive) 36 weeks + 0 days.
3. Women with singleton or multiple pregnancy.
4. Women with preterm prelabor rupture of membranes (PROM) will be included if they have uterine contractions.

Exclusion Criteria:

1. Contraindications for the use of either drugs, such as cardiac disease, hypotension, myasthenia gravis, or renal impairment.
2. Contraindications for tocolysis, such as intrauterine demise, intrauterine infection, fetal distress, placental separation, or severe pre-eclampsia.
3. Cervical dilatation > 5 cm.
4. Cervical length > 30 mm by trans-vaginal ultrasound.
5. Cervical cerclage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of women not delivered within 48 hours of starting tocolytic therapy. | 48 hours
  postponing delivery for at least 48 hours to allow the time for corticosteroid administration for fatal lung maturity

SECONDARY OUTCOMES:
Perinatal mortality | From starting treatment until 1 month of delivery
  Death of the offspring during treatment, labor or neonatal period
A composite of adverse neonatal outcomes | within 1 month of delivery
  convulsions, apnoea, asphyxia, proven meningitis, pneumothorax or sepsis
days on ventilation support | within 1 month of delivery
  number of days on mechanical ventilation
length of admission in neonatal intensive care | within 1 month of delivery
  Number of days in the NICU
Prolongation of pregnancy more than 7 days | 7 days after initiation of therapy
  Number of women not delivering after at least 7 days from starting the intervention
Delivery after 37 weeks of gestation | after 37th week of gestation
  number of women delivered after 37 weeks of gestation
Number of days till delivery | from starting the intervention until delivery
Maternal mortality rate | from starting treatment until 1 month after delivery
  Number of maternal deaths during pregnancy, labor or puerperium
Maternal infection rate | from starting treatment until 1 month after delivery
  Number of women having Chorioamnionitis, Puerperal sepsis, endometritis, or sepsis
Harm to mother from interventions (side effects) | from starting treatment until 1 month after delivery
  admission to intensive care, anaphylactic shock, dyspnoea, hypotension (leading to cardiotocography abnormalities), liver test abnormalities (elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT)), general side effects (nausea, vomiting, headache) and postpartum haemorrhage defined as >500 mL blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR